CLINICAL TRIAL: NCT03823183
Title: Protocol for a Randomized Controlled Trial With Active Control on the Effects of Combined Physical and Cognitive Training Versus Cognitive and Physical Training Separately on Executive Control and Memory Functions of Older Adults
Brief Title: Multi-domain Versus Uni-Domain Training on Executive Control and Memory Functions of Older Adults
Acronym: VIBAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: Ministry of Economy and Competitiveness (MINECO) - Government of Spain (Unknown)
Responsible Party: Principal Investigator, Soledad Ballesteros, Investigator Official Title Ph.D. Emeritus Professor of Psychology, Universidad Nacional de Educación a Distancia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: PSI2016-80377-R
Record Dates: First submitted 2019-01-07; First posted 2019-01-30 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Executive Functions; Memory Functions
Keywords: Aging, geriatrics & gerontology; Video-game cognitive training; Dance; Physical exercise; Multi-domain training; Executive functions; Memory functions; Plasticity; Transfer; Follow-up intervention; Randomized controlled trial
MeSH Terms: conditions — Motor Activity | interventions — Cognitive Training; Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: This study includes 4 intervention conditions: (1) Multi-modal Cognitive intervention + Physical intervention, (2) Cognitive intervention + Physical control, (3) Physical intervention + Cognitive control, and (4) Active Control group, Cognitive control + Physical control) x 3 (Time: Pretest, Post-test, 3-month follow-up) mixed factorial design, with "Type of training" as between-subject factors and "Time" as within-subject factor. The dependent variables will be behavioral and/or electrophysiological measures of executive functions (inhibition, shifting, working memory), memory functions (short term, episodic memory), and emotional well-being, quality of live and motivation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Multi-domain training (Experimental): Group that receives cognitive training and physical training
  Interventions: Behavioral: Cognitive training; Behavioral: Physical training
- Cognitive training (Experimental): Group that receives cognitive training and physical control activity
  Interventions: Behavioral: Cognitive training; Behavioral: Physical control
- Physical activity (Experimental): Group that receives control cognitive activity and physical training
  Interventions: Behavioral: Physical training; Behavioral: Cognitive control
- Active control (Active Comparator): Group that receives cognitive control activity and physical control activity
  Interventions: Behavioral: Cognitive control; Behavioral: Physical control

INTERVENTIONS:
Behavioral: Cognitive training — Group-based cognitive training on iPads with commercially available video games (Lumosity) designed to enhance executive control, memory functions and processing speed. Difficulty will be automatically adjusted to the performance level of the participant. Participants will train for 40 min 2 days/wk over 3 months.
  Arms: Cognitive training; Multi-domain training
Behavioral: Physical training — Group-based fitness program (senior-friendly adaption of BodyAttack) that combines aerobic, strength and coordination training to a music soundtrack. Participants will train for 40 min, 2 days/wk over 3 months.
  Arms: Multi-domain training; Physical activity
Behavioral: Cognitive control — Group-based cognitive control activity consisting of playing on iPads non-cognitively demanding video games during 40 min 2 days/wk over 3 months and exercises based on relaxation and stretching for 40 min, 2 days/wk over 3 months.
  Arms: Active control; Physical activity
Behavioral: Physical control — Group-based exercises program (based on relaxation and stretching) for 40 min, 2 days/wk over 3 months.
  Arms: Active control; Cognitive training

SUMMARY:
Age-related cognitive decline affects negatively daily living and quality of life of older adults. Previous research has shown a moderate impact of cognitive and physical training on the cognitive functioning of elders. This randomized controlled trial (RCT) examines the differential impact of multi-domain cognitive (video game training) and physical training (the physical exercise was Body-attack, a mixed of dance, aerobic, strength, and muscular resistance versus cognitive training and physical training separately, on executive control and memory functions of healthy older adults (N=120), in comparison with an active control group. Participants (between 60 and 80 years old) will be allocated randomly to one of the four experimental groups: 1) physical training-single domain: physical training and cognitive control activity; 2) cognitive training-single domain: cognitive training and physical control activity; 3) cognitive-physical multi-domain: physical training and cognitive training; 4) active control: physical control activity and cognitive control activity. Physical training will be group-based and include coordination, aerobic exercise and strength exercise. The physical control activity will include stretching and relaxation exercises. The cognitive training will consist of commercial brain training video games. Difficulty will be automatically adjusted to the performance level of the participant. The cognitive control activity will be cognitively non-demanding video games. Physical activities (experimental and control) will be trained for 40 min and cognitive activities (experimental and control) for 40 min consecutively during the same session. There will be 2 session/wk over 3 months. Executive functioning, memory functions and psychological wellbeing will be assessed using behavioral and electrophysiological measures at baseline, after study completion and at 3-month follow-up. The main goal was to investigate possible intervention-related transfer effects to untrained executive and memory functions. The goal is to find out whether multi-domain training improves more executive and memory functions that are often compromised in later years, but essential for everyday activities. We expect to find larger transfer effects in the multi-domain condition than in the uni-domain conditions, shorter ERP latencies of the P2 component, and enhanced N2 and P3b components after training.

DETAILED DESCRIPTION:
All participants complete one of the four combinations of cognitive training with video games and physical exercise. The cognitive component will be either a brain training video game program selected from Lumosity (cognitive intervention, CI) or video games not specifically designed to train attention and executive control (cognitive control, CC). The physical exercise component will be either Body-attack, a combination of dance, aerobic, strength, and muscular resistance (exercise intervention, EI) or its control condition composed of stretching, toning and relaxation (exercise control, EC).

ELIGIBILITY:
Inclusion Criteria:

No current intensive sports or physical activity practice. No current use of brain-training video games

Exclusion Criteria:

Dementia. Mild Cognitive Impairment. A neurological or major psychiatric disorder. Significant heart illness. Lung disease.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Executive functions assessed with Memory-based Task Switching | Change from Baseline in Memory-based Task Switching to 3 and 6 months
  Reaction time (RT) of correct responses in Memory-based Task Switching
Executive functions assessed with Memory-based Task Switching | Change from Baseline in Memory-based Task Switching to 3 and 6 months
  Performance in the Memory-base Task Switching: Neurophysiological parameter-Event-related potentials (ERPs) in the Memory-Based Task Switching
Attention assessed with Trail Making Test A+B | Change from Baseline in Trail Making Test to 3 and 6 months
  Performance in Trail Making Test A+B score
Inhibition assessed with Stroop Task | Change from Baseline in Stroop Task to 3 and 6 months
  Reaction time (RT) of correct responses in the Stroop Task
Working memory assessed with the N-back Task | Change from Baseline in the N-Back Task to 3 and 6 months
  Hits-False Alarms in the N-back Task
Immediate visual memory assessed with Visual Memory Face I (Weschler Memory Scale) | Change from Baseline in Face I to 3 and 6 months
  Units on the Scale: scale range (minimum score = 0 and maximum score = 48).
Differed visual memory assessed with Visual Memory Face II (Weschler Memory Scale) | Change from Baseline in Face II to 3 and 6 months
  Units on the Scale: scale range (minimum score = 0 and maximum score = 48).
  With data from Visual Memory Face I (inmediate recognition) and Visual Memory Face II (differed recognition) we compute the percentage of memory retention = Visual Memory Face II / Visual Memory Face I X 100
Immediate verbal memory assessed with Pair-Words I (Weschler Memory Scale) | Change from Baseline in Pair-Words I to 3 and 6 months
  Units on the Scale: scale range for Recall (minimum score = 0 and maximum score = 32).
Differed verbal memory assessed with Pair-Words II (Weschler Memory Scale) | Change from Baseline in Pair-Words II to 3 and 6 months
  Units on the Scale: scale range for Recall (minimum score = 0 and maximum score = 8).
  scale range for Recognition (minimum score =0 and maximum score = 24)
  Recall. With data from Pair-Words I (inmediate recognition) and Pair-Words II (differed recognition) we compute the percentage of memory retention = Pair-Words II / Pair-Word I X 100

SECONDARY OUTCOMES:
Emotional and affective wellbeing assessed with Positive and Negative Affect Schedule (PANAS) | Change from Baseline in PANAS to 3 and 6 months
  Units on the Scale: 20 items Each item is evaluated between 0 (nothing) and 5 (many). Positive emotions are assessed with items: 1, 3, 5, 7, 9, 11, 13, 15, 17, 19. Negative emotions are assessed with items: 2, 4, 6, 8, 10, 12, 14, 16, 18, 20.
Emotional and affective wellbeing assessed with The Life Satisfaction Index (LSI): 20 items Each item is assessed using two-point agree/disagree score rated items 0 for a response indicating dissatisfaction and 1 for satisfaction. | Change from Baseline in LSI to 3 and 6 months
  Units on the Scale: 20 items A two-point agree/disagree score rated items 0 for a response indicating dissatisfaction and 1 for satisfaction.
Cardio-respiratory capacity assessed with the 6 Minutes Walk Test | Change from Baseline in 6 Minutes Walk Test to 3 and 6 months
  Physiological parameter
Physical dimension assessed with The Short Physical Performance Battery (SPPB) | Change from Baseline in SPPB to 3 and 6 months
  Units on the Scale
Demographic interview and medical history | Baseline
  Respond to questions related to demographics and medical history
General cognitive state assessed with Mini Mental State Examination (MMSE) | Baseline
  Units on the test: scale range (minimum score = 0 and maximum score = 30). Values between 27 and 30 points are considered as "appropriate cognitive state".
  Values between 24 and 26 points are considered as "possible mild cognitive impairment" Values between 0 and 23 points are considered as "possible dementia". This test is a screening test and it is not adequate to diagnose. In this protocol participants with scores under 27 will be excluded from the study.
General depression state assessed with Yesavage Abbreviate Questionnaire. (GDS) | Baseline
  Units on the test: scale range (minimum score = 0 and maximum score = 15). Values between 0 and 5 points are considered as "no depression". Values between 5 and 10 points are considered as "mild depression" Values between 10 and 15 points are considered as "severe depression". This test is a screening test and it is not adequate to diagnose. In this protocol participants with scores greater than 5 will be excluded from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Ballesteros, PhD, Principal Investigator — UNED
Locations (1):
- Department of Basic Psychology II (UNED), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ballesteros S, Rieker JA, Mayas J, Prieto A, Toril P, Jimenez MP, Reales JM. Effects of multidomain versus single-domain training on executive control and memory in older adults: study protocol for a randomized controlled trial. Trials. 2020 May 14;21(1):404. doi: 10.1186/s13063-020-04293-3. PMID 32410715